CLINICAL TRIAL: NCT05052918
Title: The Effect of Exercise and Metformin on Carotid Intima-media Thickness in Patients With Prediabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXERCISECIMT
Record Dates: First submitted 2021-09-07; First posted 2021-09-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Pre Diabetes; Exercise; Metformin; Atherosclerosis
Keywords: Prediabetes; exercise; metformin; atherosclerosis
MeSH Terms: conditions — Glucose Intolerance; Motor Activity; Atherosclerosis; Prediabetic State | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercise (Active Comparator): Patients with prediabetes undergoing a 12-week exercise program
  (1 hour of moderate-intensity aerobic exercise 3 days a week for 12 weeks)
  Interventions: Behavioral: Exercise
- Control (No Intervention): Patients with prediabetes with no intervention
- Metformin (No Intervention): Patients with prediabetes using metformin

INTERVENTIONS:
Behavioral: Exercise — 1 hour of moderate-intensity aerobic exercise 3 days a week for 12 weeks
  Arms: Exercise

SUMMARY:
The aim of this study is to evaluate whether there is a change in carotid intima media thickness with the application of guide-based exercise programs in individuals with prediabetes, and to evaluate whether there is a difference between the group in which exercise programs were applied and those who received only lifestyle change and metformin.

DETAILED DESCRIPTION:
The researchers think that the application of guide-based exercise programs in prediabetes patients will decrease the carotid intima-media thickness.The aim of this study is to evaluate whether there is a change in carotid intima media thickness with the application of guide-based exercise programs in individuals with prediabetes, and to evaluate whether there is a difference between the group in which exercise programs were applied and those who received only lifestyle change and metformin.

ELIGIBILITY:
Inclusion Criteria:

* Leading a sedentary life
* Those who have sufficient motivation to participate in the exercise program (will be evaluated by a one-on-one interview by the researchers)
* Have the same weight for 6 months before participating in the study (±2.5 kg)
* Those diagnosed with prediabetes by oral glucose tolerance test and/or HbA1c measurement

Exclusion Criteria:

* Serious medical condition (for example, advanced malignancy or major neurological, psychiatric or endocrine disease, respiratory failure, etc.) that would prevent the person from participating in exercise training.
* Having cardiovascular disease
* Being diabetic
* Using metformin before participating in the study
* Receiving hormone replacement therapy
* Life expectancy less than 1 year
* HIV positivity
* Substance use
* Functional dependency
* Cognitive weakness
* Those who have other diseases that will affect the results of the study (respiratory diseases, muscle diseases, etc.)
* Those who use drugs or supplements that will affect the results of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-08 (Actual); Primary Completion 2023-03-15 (Estimated); Study Completion 2023-03-15 (Estimated)

PRIMARY OUTCOMES:
Carotid ultrasound | 12 weeks
  milimeter size of carotid intima media thickness

CONTACTS AND LOCATIONS:
Overall Officials: Elif Yıldırım Ayaz, M.D., Principal Investigator — Sultan Abdülhamid Han Training and Research Hospital
Locations (1):
- Sultan Abdülhamid Han Training and Research Hospital, Üsküdar, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided